CLINICAL TRIAL: NCT01288196
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Immunogenicity of CNTO 6785 Following a Single Intravenous or a Single Subcutaneous Administration in Healthy Subjects
Brief Title: A Safety, Tolerability, Pharmacokinetics, and Immunogenicity Study of CNTO 6785 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017752; CNTO6785OPD1001
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: CNTO 6785; Intravenous; Subcutaneous; Pharmacokinetics; Immunogenicity; Safety; Tolerability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- 001 (Experimental): CNTO 6785 1 mg/kg IV A single 30-minute IV infusion of CNTO 6785 1 mg/kg
  Interventions: Drug: CNTO 6785 1 mg/kg IV
- 002 (Experimental): CNTO 6785 3 mg/kg IV A single 30-minute IV infusion of CNTO 6785 3 mg/kg
  Interventions: Drug: CNTO 6785 3 mg/kg IV
- 003 (Experimental): CNTO 6785 10 mg/kg IV A single 30-minute IV infusion of CNTO 6785 10 mg/kg
  Interventions: Drug: CNTO 6785 10 mg/kg IV
- 004 (Placebo Comparator): Placebo IV A single 30-minute IV infusion of placebo
  Interventions: Drug: Placebo IV
- 005 (Experimental): CNTO 6785 SC A single SC dose of CNTO 6785 (3 mg/kg) administered in up to 3 SC injections
  Interventions: Drug: CNTO 6785 SC
- 006 (Placebo Comparator): Placebo SC A single SC dose of placebo administered in up to 3 SC injections
  Interventions: Drug: Placebo SC

INTERVENTIONS:
Drug: Placebo IV — A single 30-minute IV infusion of placebo
  Arms: 004
Drug: CNTO 6785 1 mg/kg IV — A single 30-minute IV infusion of CNTO 6785 1 mg/kg
  Arms: 001
Drug: CNTO 6785 3 mg/kg IV — A single 30-minute IV infusion of CNTO 6785 3 mg/kg
  Arms: 002
Drug: CNTO 6785 10 mg/kg IV — A single 30-minute IV infusion of CNTO 6785 10 mg/kg
  Arms: 003
Drug: CNTO 6785 SC — A single SC dose of CNTO 6785 (3 mg/kg) administered in up to 3 SC injections
  Arms: 005
Drug: Placebo SC — A single SC dose of placebo administered in up to 3 SC injections
  Arms: 006

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, blood levels, and immune responses of CNTO 6785 after administration to healthy adult volunteers.

DETAILED DESCRIPTION:
This is a randomized (study drug will be assigned by chance), double-blind (neither the volunteer, physician, or study staff will know the identity of the assigned treatment), study to evaluate the safety, tolerability, pharmacokinetics (blood levels of drug) and immunogenicity (development of antibodies to the drug) of a single dose of CNTO 6785 administered to healthy adult volunteers intravenously (in the vein) or by subcutaneous (under the skin) administration to healthy adult volunteers.This will be the first administration of CNTO 6785 to humans; therefore, no clinical experience is available. Healthy volunteers will receive a single dose of 1, 3, or 10 mg/kg of CNTO 6785 or placebo as a 30-minute intravenous (IV) (injection into a blood vessel) infusion or a single dose of 3 mg/kg of CNTO 6785 administered in up to 3 subcutaneous (under the skin) (SC) injections.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteer with no clinically significant abnormalities as determined by the investigator (study physician)
* Have a body mass index (BMI) between 19-30 kg/m2
* Be a non-smoker for at least 6 months prior to study participation
* Women must be postmenopausal or surgically sterile

Exclusion Criteria:

* Currently have or have a history of any clinically significant medical illness or medical disorders (includes malignancies or serious infections) that the investigator (study physician) considers should exclude the volunteer from the study
* Major surgery or significant trauma within 12 weeks of screening
* Any volunteer who plans to undergo elective surgery within 4 weeks prior to study agent administration and through the end of the study
* Consumes, on average, more than approximately 500 mg/day of caffeine (as contained in 5 cups of tea or coffee or 8 cans of soda or other caffeinated products per day).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number and type of adverse events reported | Up to Week 17
Number and type of Infusion (injection) site reactions | Up to Week 17
Vital signs measurements | Up to Week 17
Clinical laboratory test results | Up to Week 17
Findings from cardiology assessments (electrocardiograms [ECGs] and cardiac telemetry) | Up to Week 17

SECONDARY OUTCOMES:
Serum concentration of CNTO 6785 | Up to Week 17
Serum antibodies to CNTO 6785 | Up to Week 17

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Merksem, Belgium